CLINICAL TRIAL: NCT02089113
Title: A Prospective, Multicenter, Randomized, Parallel-Arm, Double-Masked, Vehicle Controlled Phase 3B Study Evaluating the Safety and Efficacy of OTX-DP for the Treatment of Ocular Inflammation and Pain After Cataract Surgery
Brief Title: OTX-14-003: A Phase 3 Study Evaluating the Safety and Efficacy of OTX-DP for the Treatment of Ocular Inflammation and Pain After Cataract Surgery
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ocular Therapeutix, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: OTX-14-003
Record Dates: First submitted 2014-03-13; First posted 2014-03-17 (Estimated); Results first posted 2016-03-30 (Estimated); Last update posted 2019-09-26 (Actual); Status verified 2019-09

CONDITIONS: Post-Surgical Ocular Pain; Post-Surgical Ocular Inflammation
MeSH Terms: interventions — Dexamethasone

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- OTX-DP (Experimental): OTX-DP (dexamethasone insert) 0.4 mg for intracanalicular use
  Interventions: Drug: Dexamethasone
- PV (Placebo Comparator): PV (placebo drug delivery vehicle)
  Interventions: Procedure: Placebo Vehicle

INTERVENTIONS:
Drug: Dexamethasone
  Arms: OTX-DP
Procedure: Placebo Vehicle
  Arms: PV

SUMMARY:
The objective of the study was to evaluate the safety and efficacy of OTX-DP (dexamethasone insert) 0.4 mg for intracanalicular use when placed in the canaliculus of the eyelid for the treatment of post-surgical inflammation and pain in subjects who had undergone cataract extraction with intraocular lens implantation

ELIGIBILITY:
Inclusion Criteria:

* Has a cataract and is expected to undergo clear corneal cataract surgery with phacoemulsification and implantation of a posterior chamber lens
* Has a potential post-operative pinhole corrected Snellen VA of at least 20/200 or better in both eyes

Exclusion Criteria:

* Any intraocular inflammation in the study eye present during the screening slit lamp examination
* Score greater than "0" on the Ocular Pain Assessment in the study eye at Screening
* Any intraocular inflammation in the study eye present during the screening slit lamp examination

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 241 (Actual)
Dates: Start 2014-04 (Actual); Primary Completion 2015-01 (Actual); Study Completion 2015-03 (Actual)

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Dexamethasone Punctum Plug: Drug treatment
- Placebo Vehicle Punctum Plug: No drug treatment
Period: Overall Study
Arm/Group | Dexamethasone Punctum Plug | Placebo Vehicle Punctum Plug
Started | 161 | 80
Completed | 160 | 80
Not Completed | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- OTX-DP (Dexamethasone Punctum Plug): Resorbable hydrogel drug delivery vehicle containing dexamethasone
  Dexamethasone
- PVPP (Placebo Punctum Plug): Resorbable hydrogel drug delivery vehicle containing no drug
  Punctum Plug
- Total: Total of all reporting groups
Arm/Group | OTX-DP (Dexamethasone Punctum Plug) | PVPP (Placebo Punctum Plug) | Total
Number analyzed (Participants) | 161 | 80 | 241
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 49 | 22 | 71
  >=65 years | 112 | 58 | 170
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 98 | 39 | 137
  Male | 63 | 41 | 104

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With an Absence of Anterior Chamber Inflammation
Description: Absence of cells (i.e., score of '0') in the anterior chamber of the study eye at Day 14
Time Frame: Day 14
Measure: Number; unit: participants
Groups:
- Placebo Vehicle: PV (placebo drug delivery vehicle)
Arm/Group | OTX-DP | Placebo Vehicle
Number analyzed (Participants) | 161 | 80
participants | 63 | 25

2. Primary Outcome: Number of Participants With an Absence of Ocular Pain
Description: Absence of pain (i.e., score of '0') in the study eye at Day 8
Time Frame: Day 8
Measure: Number; unit: participants
Arm/Group | OTX-DP | Placebo Vehicle
Number analyzed (Participants) | 161 | 80
participants | 124 | 47

ADVERSE EVENTS:
Arm/Group | Dexamethasone Punctum Plug | Placebo Vehicle Punctum Plug
Serious Adverse Events (participants affected / at risk) | 0/160 | 1/80
Other Adverse Events (participants affected / at risk) | 0/160 | 0/80
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dexamethasone Punctum Plug (N=160) | Placebo Vehicle Punctum Plug (N=80)
mental disorder (Psychiatric disorders) | 0 | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No